CLINICAL TRIAL: NCT05308420
Title: Pericapsular Nerve Group (PENG) Block vs Intrathecal Morphine for Postoperative Analgesia in Patients Undergoing Total Hip Arthroplasty: a Randomized Non-inferiority Trial
Brief Title: PENG Block vs Intrathecal Morphine in Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kresimir Oremus, MD (Other)
Responsible Party: Sponsor-Investigator, Kresimir Oremus, MD, Head of Division of Anesthesiology, Akromion Special Hospital for Orthopedic Surgery
Organization: Akromion Special Hospital for Orthopedic Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 022021
Record Dates: First submitted 2022-03-18; First posted 2022-04-04 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Total Hip Arthroplasty; Postoperative Pain
Keywords: Total hip arthroplasty; Postoperative pain; Anesthesia, Regional
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion; Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: Non-inferiority randomized triple-blinded controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization and study drug preparation by person(s) not involved in patient care, data gathering or outcome evaluation. Group allocation kept in sealed opaque envelope until all data gathered. Outcome assessor/statistician will be blinded as to which group received which intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block (Active Comparator): Patients scheduled for primary total hip arthroplasty after receiving spinal anesthesia will undergo pericapsular nerve group (PENG) block.
  Postoperative multimodal analgesia with paracetamol, etoricoxib and oxycodone
  Interventions: Procedure: Pericapsular nerve group (PENG) block; Procedure: Spinal anesthesia; Drug: Intrathecal placebo
- Intrathecal morphine (Active Comparator): Patients scheduled for primary total hip arthroplasty will receive spinal anesthesia with local anesthetic and morphine administered intrathecally. After onset of spinal anesthesia a sham PENG block will be performed.
  Postoperative multimodal analgesia with paracetamol, etoricoxib and oxycodone.
  Interventions: Procedure: Spinal anesthesia; Drug: Intrathecal morphine; Procedure: Sham PENG block

INTERVENTIONS:
Procedure: Pericapsular nerve group (PENG) block — A 22 gauge 120mm nerve block needle will be introduced under ultrasound guidance in plane from superolateral to posteromedial to position the needle tip posterolateral to the ileopsoas tendon in-between the anterior inferior iliac spine and the ileopubic (ileopectineal) eminence and 20ml 0.5% levobupivacaine with 2mg (0.5ml) dexamethasone injected (total volume of injectate 20.5ml) between the tendon and the inferior pubic ramus just proximal to the attachment of the anterior hip capsule
  Arms: PENG block
Procedure: Spinal anesthesia — Spinal anesthesia will be performed at the level of the presumed interspace in-between the third and fourth lumbar vertebrae by introducing a 27 gauge pencil-point spinal needle and 15mg of levobupivacaine (3ml) injected intrathecally
Drug: Intrathecal morphine — 100 micrograms of preservative free morphine diluted to a volume of 0.5ml is added to the local anesthetic solution injected for spinal anesthesia (total injectate volume 3.5ml)
  Arms: Intrathecal morphine
Procedure: Sham PENG block — A 22 gauge 120mm nerve block needle will be introduced under ultrasound guidance in plane from superolateral to posteromedial to position the needle tip posterolateral to the ileopsoas tendon in-between the anterior inferior iliac spine and the ileopubic (ileopectineal) eminence and a placebo solution consisting of 20.5ml 0.9%NaCl injected between the tendon and the inferior pubic ramus just proximal to the attachment of the anterior hip capsule
  Arms: Intrathecal morphine
Drug: Intrathecal placebo — 0.5ml of placebo solution (0.9%NaCl) is added to the local anesthetic solution injected for spinal anesthesia (total injectate volume 3.5ml)
  Arms: PENG block

SUMMARY:
To compare the impact of pericapsular nerve group (PENG) block to intrathecal morphine on postoperative analgesia, motor function and side effects in patients undergoing primary total hip arthroplasty under spinal anesthesia.

DETAILED DESCRIPTION:
The study aims to confirm the non-inferiority of PENG block vs intrathecal morphine in patients undergoing total hip arthroplasty under spinal anesthesia. Non-inferiority will be assessed regarding maximum pain on a numerical rating scale at rest and during active hip flexion and regarding cumulative morphine consumption during 48 postoperative hours. Impact on quadriceps muscle motor function and side effects including pruritus, nausea and vomiting and hypotension will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with osteoarthritis of the hip scheduled for primary total hip arthroplasty under spinal anesthesia able to provide written informed consent

Exclusion Criteria:

* patient unwilling / unable to provide informed consent
* contraindications for any of the drugs and procedures included in the study protocol (allergies, local infection, coagulopathy)
* high risk for perioperative morbidity/mortality (ASA Physical Status Classification IV)
* preoperative use of strong opioid analgesia (due to hip pain or other acute/chronic pain condition)
* pregnancy
* substance abuse

Post Randomization Exclusion Criteria:

* change of surgical plan
* violation of study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-03 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Maximum pain at rest | 48 postoperative hours
  maximum pain on a numerical rating scale at rest over first 48 post-operative hours Test treatment (PENG block) is to be considered non-inferior to reference treatment (intrathecal morphine) only if during final data analysis conditions of non-inferiority are met for all 3 co-primary outcomes
Maximum pain with active hip flexion | 48 postoperative hours
  maximum pain on a numerical rating scale with active 60 degrees hip flexion over first 48 post-operative hours Test treatment (PENG block) is to be considered non-inferior to reference treatment (intrathecal morphine) only if during final data analysis conditions of non-inferiority are met for all 3 co-primary outcomes
cumulative morphine equivalent dose over 48 post-operative hours | 48 postoperative hours
  cumulative opioid consumption including morphine rescue analgesia will be recorded during the first 48 postoperative hours Test treatment (PENG block) is to be considered non-inferior to reference treatment (intrathecal morphine) only if during final data analysis conditions of non-inferiority are met for all 3 co-primary outcomes

SECONDARY OUTCOMES:
Quadriceps muscle motor block | 24 postoperative hours
  Quadriceps muscle motor function will be evaluated by a straight leg raise test performed at 4,6,12,20 and 24 hours postoperatively
Opioid side effects | 48 postoperative hours
  The presence of pruritus, nausea and vomiting, hypotension and need for rescue antiemetic medication (ondansetron) will be monitored and recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Akromion Special Hospital for Orthopedic Surgery, Krapinske Toplice, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Hess SR, Lahaye LA, Waligora AC, Sima AP, Jiranek WA, Golladay GJ. Safety and side-effect profile of intrathecal morphine in a diverse patient population undergoing total knee and hip arthroplasty. Eur J Orthop Surg Traumatol. 2019 Jan;29(1):125-129. doi: 10.1007/s00590-018-2293-9. Epub 2018 Aug 13. PMID 30105593
- [Background] Anger M, Valovska T, Beloeil H, Lirk P, Joshi GP, Van de Velde M, Raeder J; PROSPECT Working Group* and the European Society of Regional Anaesthesia and Pain Therapy. PROSPECT guideline for total hip arthroplasty: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 Aug;76(8):1082-1097. doi: 10.1111/anae.15498. Epub 2021 May 20. PMID 34015859
- [Derived] Oremus K, Trkulja V, Gasparini G, Sostaric S, Cicak N, Haspl M, Mihaljevic S. Pericapsular nerve group (PENG) block compared to intrathecal morphine for analgesic efficacy in total hip arthroplasty: A placebo-controlled randomized double-blind non-inferiority trial. J Clin Anesth. 2025 Sep;106:111921. doi: 10.1016/j.jclinane.2025.111921. Epub 2025 Jul 2. PMID 40609218